CLINICAL TRIAL: NCT06684730
Title: Comparison of Standard Myoelectric Hand and Bionic Hand Use in Individuals With Upper Limb Amputation
Status: Recruiting | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nurdan Korkmaz, Physical Medicine and Rehabilitation Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: E-34215015-771-250527790
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Transradial Amputation; Wrist Disarticulation
Keywords: Standard Myoelectric Hand; Transradial Amputation; Bionic Hand; Wrist disarticulation; Amputation of upper limb

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with transradial amputees or wrist disarticulation using standard myoelectric hands
  Interventions: Procedure: Hand Function Assessment Scales; Other: Prosthesis Satisfaction Scale; Other: Quality of Life Scale; Procedure: Kinematic Analysis; Procedure: Parkour Completion Time; Procedure: Fatigue Scale
- Individuals with transradial amputees or wrist disarticulation using bionic hand
  Interventions: Procedure: Hand Function Assessment Scales; Other: Prosthesis Satisfaction Scale; Other: Quality of Life Scale; Procedure: Kinematic Analysis; Procedure: Parkour Completion Time; Procedure: Fatigue Scale

INTERVENTIONS:
Procedure: Hand Function Assessment Scales — The Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH), The Box and Block Test (BBT) and Action Research Arm Test (ARAT) will be used as hand function assessment scales.
Other: Prosthesis Satisfaction Scale — The Quebec Assistive Technology User Satisfaction Assessment (Q-YTKMD) Questionnaire will be used.
Other: Quality of Life Scale — 5Q-5D-5L will be used as quality of life scale.
Procedure: Kinematic Analysis — Kinematic analysis of shoulder abduction, elbow flexion, and cervical flexion will be performed during simulated tasks of drinking water from a glass and filling glass of water.
Procedure: Parkour Completion Time — A 10-item daily living activities parkour will be prepared for the participants. During the parkour, the participant will be given the following tasks: opening and closing 10 jar lids, slicing a 20cm cylindrical dough into 10 pieces, simulating drinking soup from a bowl 15 times with a spoon (standard bowl 150 ml, standard tablespoon 10 ml), simulating eating meatballs from a plate with a fork 10 times (approximately 6-10 meatballs per serving), simulating pouring water from a pitcher into a glass 10 times, simulating drinking water from a glass 10 times, simulating brushing teeth for 2 minutes, opening 10 clothespins attached to the edge of a cardboard box and attaching them to the other side, simulating opening and closing a zipper, and putting on shoes and tying shoelaces. The course completion time will be recorded.
Procedure: Fatigue Scale — A pre- and post-parkour will be employed, including a 5-point Likert scale for fatigue assesment, hand function assessment scales and kinematic analysis to participants. The results before and after the parkour will be compared.

SUMMARY:
This single-center, prospective, comparative study aims to compare hand function, quality of life, patient satisfaction, task completion time, fatigue, and compensatory elbow, shoulder, and cervical movements in individuals with transradial amputation or wrist disarticulation who use either standard myoelectric or bionic hand prostheses. The primary research questions are:

1. Are there differences in patient satisfaction, quality of life, and hand function between individuals using standard myoelectric and bionic hand prostheses?
2. Do individuals using standard myoelectric and bionic hand prostheses exhibit different kinematics in terms of compensatory shoulder, elbow, and neck movements? Could bionic hand prostheses with their diverse grasping capabilities lead to fewer compensatory movements compared to standard myoelectric hand prostheses?
3. Can fatigue induced by performing specific activities of daily living alter hand function and upper extremity-neck kinematics in individuals using either standard myoelectric or bionic hand prostheses?
4. Can cognitive and physical fatigue following activities of daily living lead to different levels of changes in hand function and upper extremity-neck kinematics in individuals using standard myoelectric and bionic hand prostheses?

DETAILED DESCRIPTION:
Amputation constitutes a major trauma that substantially affects an individual's functional status and activities of daily living. The functional impairments ensuing from amputation can impede reintegration into normal life, giving rise to social, occupational, and psychological challenges. Amputees frequently encounter significant limitations in activities and participation. These limitations are predominantly related to mobility and self-care. These factors adversely affect the ability to return to work and maintain employment, continue social relationships, engage in leisure pursuits, and be active in community life. A variety of prostheses are employed to restore the functions of an amputated limb and achieve bodily integrity. Individuals with upper limb amputations may utilize cosmetic (passive), body-powered (mechanical, cable-activated), myoelectric, or hybrid prostheses. Myoelectric prostheses are controlled by electromyography (EMG) signals and are powered by rechargeable motors to execute movements. Successful prosthesis use necessitates the individual's physical capacity to operate the device and sufficient cognitive awareness to comprehend and control it. Two prevalent hand types in myoelectric upper limb prostheses are the standard myoelectric hand and the bionic hand. The standard myoelectric hand employs a single motor to provide a robust and consistent tripod grasp. The motor actuates the opening and closing of the first, second, and third digits. The fourth and fifth digits passively follow the others. Bionic hands, in contrast, feature multiple joints in each finger, enabling more natural finger movements, and some models incorporate multiple motors for independent finger control. This expands the range of functional grasp patterns. Instead of a single tripod grasp, they offer various grasp patterns (pinch, trigger, lateral, cylindrical, spherical, hook, key grasp, etc.). While providing users with greater hand dexterity, this increased grasp versatility comes with drawbacks such as higher cost and reduced durability. Moreover, the sequential nature of grasp movements, the necessity for patients to memorize this sequence, and the need to switch modes between grasps (open, dual, triple, co-contraction, button) can pose usability challenges. Consequently, executing a hand function using these grasps can be time-consuming, cognitively demanding, and physically exhausting. Despite over a decade of use, the existing literature on the advantages and disadvantages of bionic hand prostheses is limited and the findings are not entirely compelling. Additionally, these few studies predominantly rely on user reports. Individuals with upper limb amputation who use prostheses demonstrate unnatural or unusual movements in other joints and body regions. To successfully perform activities of daily living and tasks, they adapt the movement of their remaining limbs and develop compensatory movements. As the prosthesis's functionality approaches that of a healthy hand, compensatory movements also diminish. Studies have shown that during the use of upper limb prostheses, shoulder and trunk joint angles are increased compared to healthy individuals, elbow range of motion is limited, and decreased elbow movement is compensated for by increasing shoulder abduction or cervical spine flexion. These compensatory movements result in cognitive and physical fatigue in amputees. This situation is considered one of the factors influencing the discontinuation of prosthesis use. While the literature suggests that the use of bionic hands may reduce these compensatory movements, only one study has compared these angles in individuals using standard myoelectric hands and bionic hands. To our knowledge, there is no study that comprehensively compares quality of life, prosthesis satisfaction, kinematic measurement of compensatory elbow, shoulder, and cervical movements, time-consuming of hand functions, and the degree of fatigue in individuals with upper limb amputation who use bionic or standard myoelectric hands. This study aims to address this gap in the literature, evaluate the functionality of prostheses more objectively by combining various outcome measures, and to pioneer new studies.

ELIGIBILITY:
Inclusion Criteria:

* Having a transradial amputation or wrist disarticulation due to acquired or congenital causes,
* Using a standard myoelectric or bionic hand prosthesis for at least 6 months,
* Being between the ages of 18 and 65,
* Having no neurological or cognitive disorders, rheumatic diseases, or other upper extremity dysfunction that could affect test results, and
* Having signed an informed consent form indicating the patient's willingness to participate in the study.

Exclusion Criteria:

* Individuals younger than 18 or older than 65,
* Those with additional musculoskeletal or neurological conditions preventing them from completing the tests and scales,
* Those with psychiatric disorders or cognitive impairments preventing them from completing the questionnaire and assessment scales,
* Those with stump or upper extremity conditions preventing them from using their prosthesis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-two participants with transradial amputation or wrist disarticulation will be enrolled in the study. These participants will be recruited from the Veterans Physical Therapy and Rehabilitation Training and Research Hospital and will consist of 11 individuals using bionic hand prostheses and 11 using standard myoelectric hand prostheses.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-11-27 (Estimated); Primary Completion 2025-08-27 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Kinematical measurement of shoulder abduction | immediately before/after the parkour
  Kinovea, a free and reliable 2D motion analysis software, will be used to collect kinematic data during simulated tasks of pouring water from a pitcher into a glass and drinking water from an empty glass. Kinovea provides acceptable accuracy in angular and linear measurements obtained by digitizing x and y coordinates. In the study, two synchronized cameras will be positioned 150 cm away from the patient, anteriorly and laterally, to capture the lumbar region and more proximal segments. Markers will be placed on the lateral epicondyle and fossa cubitalis of the elbow, and on the anterior and lateral aspects of the glenohumeral joint. Shoulder abduction kinematics will be assessed.

SECONDARY OUTCOMES:
Defined parkour completion time | From the start of the parkour to the completion of the parkour (about 12 minutes)
  A 10-item daily living activities parkour will be prepared for the participants. During the parkour, the participant will be given the following tasks: opening and closing 10 jar lids, slicing a 20cm cylindrical dough into 10 pieces, simulating drinking soup from a bowl 15 times with a spoon (standard bowl 150 ml, standard tablespoon 10 ml), simulating eating meatballs from a plate with a fork 10 times (approximately 6-10 meatballs per serving), simulating pouring water from a pitcher into a glass 10 times, simulating drinking water from a glass 10 times, simulating brushing teeth for 2 minutes, opening 10 clothespins attached to the edge of a cardboard box and attaching them to the other side, simulating opening and closing a zipper, and putting on shoes and tying shoelaces. The course completion time will be recorded.
The Box and Blocks Test (BBT) | "Immediately before/after parkour
  The Box and Blocks Test (BBT) is a standardized assessment of unimanual dexterity. It involves transferring 150 cubic wooden blocks, one at a time, from one compartment of a divided wooden box to the other within a one-minute time limit. The test score is determined by the total number of blocks transferred, with higher scores indicating greater dexterity.
Action Research Arm Test (ARAT) | Immediately before/after parkour
  The Action Research Arm Test (ARAT) is a standardized 19-item assessment designed to evaluate upper limb function. Tasks are hierarchically arranged from complex to simple and are categorized into four subscales: gross grasp, fine grasp, pinch, and gross movement. A 4-point ordinal scale, ranging from 0 (no movement) to 3 (normal movement), is used to score each item. Total scores range from 0 to 57, with higher scores indicating better upper limb function.
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | Immediately before/after parkour
  This is a commonly used 30-item outcome assessment tool designed to quantify the physical, psychological, and social role function in individuals experiencing upper extremity dysfunction. The questionnaire employs a 5-point Likert scale for scoring, where a higher score signifies a more pronounced level of disability.
Kinematic measurement of elbow flexion | Immediately before/after parkour
  Kinovea software will be used during simulated tasks of pouring water from a pitcher into a glass and drinking water from an empty glass. Two synchronized cameras will be positioned 150 cm away from the patient, anteriorly and laterally, to capture the lumbar region and more proximal segments. Markers will be placed on the lateral epicondyle and fossa cubitalis of the elbow, anteriorly and laterally on the glenohumeral joint, and on the dorsal aspect of the hand. Elbow flexion kinematics will be evaluated.
Kinematic measurement of cervical flexion | Immediately before/after parkour
  Kinovea software will be used during simulated tasks of pouring water from a pitcher into a glass and drinking water from an empty glass. Two synchronized cameras will be positioned 150 cm away from the patient, anteriorly and laterally, to capture the lumbar region and more proximal segments. Markers will be placed on the C7 vertebra and the occiput. Cervical flexion kinematics will be evaluated.
5Q-5D-5L | Baseline
  The 5Q-5D-5L is a generic quality of life scale. The scale is divided into two sections. The first section assesses the daily health profile in five sub-dimensions: movement, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents rate each sub-dimension on a 5-point Likert scale ranging from "no problem" to "extreme problem". In the second section, participants rate their current health status on a 0-100 scale, marking their response on a thermometer-like scale.
The Quebec Assistive Technology User Satisfaction Assessment (Q-YTKMD) Questionnaire | Baseline
  The Q-YTKMD questionnaire is a standardized tool commonly used to evaluate the satisfaction of individuals using a variety of assistive technologies. It comprises 12 items, specifically addressing satisfaction with the assistive device (8 items) and the service provided (4 items). Scores range between 12 and 60, with higher scores reflecting greater levels of satisfaction.
Fatigue Assessment Scale | Immediately before/after parkour
  It is a 5-point Likert scale ranging from 0 (not tired at all) to 5 (very tired).

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Therapy and Rehabilitation Training and Research Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Major MJ, Stine RL, Heckathorne CW, Fatone S, Gard SA. Comparison of range-of-motion and variability in upper body movements between transradial prosthesis users and able-bodied controls when executing goal-oriented tasks. J Neuroeng Rehabil. 2014 Sep 6;11:132. doi: 10.1186/1743-0003-11-132. PMID 25192744
- [Background] Carey SL, Dubey RV, Bauer GS, Highsmith MJ. Kinematic comparison of myoelectric and body powered prostheses while performing common activities. Prosthet Orthot Int. 2009 Jun;33(2):179-86. doi: 10.1080/03093640802613229. PMID 19367522
- [Background] Kerver N, Schuurmans V, van der Sluis CK, Bongers RM. The multi-grip and standard myoelectric hand prosthesis compared: does the multi-grip hand live up to its promise? J Neuroeng Rehabil. 2023 Feb 15;20(1):22. doi: 10.1186/s12984-023-01131-w. PMID 36793049